CLINICAL TRIAL: NCT00853437
Title: Comparison of Techniques for Assessing Cardiac Output and Preload in Critically Ill Pediatric Patients
Acronym: GCH
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-COSTATUS-2A-H; 2R44HL061994-04A2 (NIH)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output
Keywords: Comparison of CO by new method to clinician's estimate and implied CO from the measurement of arteriovenous oxygen content difference.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The ability to measure cardiac output (CO) accurately and reproducibly at frequent intervals remains elusive to the clinician caring for critically ill pediatric patients even though a large proportion of these children are known to have hemodynamic compromise as a result of their illness. Current techniques used in adults to measure CO are not suitable for routine use with pediatric patients. A new ultrasound dilution approach provides an opportunity to measure cardiac output and blood volumes in pediatric patients. The main aim of this study is to compare CO measured by the new method with the clinician's estimate and implied CO from the measurement of the arteriovenous oxygen content difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients with in situ central venous and arterial catheters
* Ability to draw blood from arterial and central venous catheters
* Presence of parent or guardian to provide consent

Exclusion Criteria:

* Patients over 16 years of age.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (up to 16 years of age ) in the ICU with in situ central venous and arterial catheters.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Compare CO measured by the new method with clinician's estimate and implied CO from measurement of arteriovenous oxygen content difference. | 5-8 minutes minimum

SECONDARY OUTCOMES:
Measure blood volumes to compare effects of volume infusion and furosemide. | 5-8 minutes minimum

CONTACTS AND LOCATIONS:
Overall Officials: Karen Powers, MD, Principal Investigator — Golisano Children's Hospital
Locations (1):
- Golisano Children's Hospital, Rochester, New York, United States

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416